CLINICAL TRIAL: NCT02734472
Title: Effect of the Interaction Between Environmental Factors and Genetic Predisposition on Long-term Blood Pressure in Chinese Population
Brief Title: Blood Pressure Follow-up Study in Two Chinese Cohorts(C-BPCS)
Acronym: C-BPCS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF-CRF-2015-006
Record Dates: First submitted 2016-03-22; First posted 2016-04-12 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Hypertension
Keywords: blood pressure; Hypertrophy, Left Ventricular; Vascular Stiffness; Proteinuria; Carotid Artery Diseases
MeSH Terms: conditions — Hypertension; Hypertrophy, Left Ventricular; Proteinuria; Carotid Artery Diseases | interventions — Incidence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Meixian county adult salt-sensitive hypertension study is a family-based dietary interventional study. Whole blood specimen was collected from each participant who underwent a chronic salt load and potassium supplementation trial.Genomic DNA was extracted from whole blood specimen using the GOLDMAG Whole Blood Genomic DNA Purification Kit.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Hanzhong cohort: A total of 4623 adolescents aged 6-15 years old in Hanzhong rural areas were recruited in 1987.During the follow-up period, the information about the incidence and risk factors of hypertension will be collected.
  Interventions: Other: Incidence and risk factors of hypertension
- Mei county cohort: A total of 675 individuals from 126 families were recruited in this family-based dietary intervention study. A community-based BP screening was conducted among adults aged 18-60 years in the study villages. The probands who had a mean systolic BP (SBP) between 130-160 mmHg and/or a diastolic BP (DBP) between 85-100 mmHg and no use of antihypertensive medications and their parents, siblings, spouses, and offspring were recruited in this study. During the follow-up period, the information about the incidence and risk factors of hypertension will be collected.
  Interventions: Other: Incidence and risk factors of hypertension

INTERVENTIONS:
Other: Incidence and risk factors of hypertension — During the follow-up period,General information(age, sex, BMI, blood pressure, the history of drink and smoke, medical history, etc).Blood biochemistry parameters（Lipid, hsCRP levels, etc）and other laboratory examination parameters(arterial stiffness,IMT, FMD) will be collected.

SUMMARY:
Essential hypertension is a complex trait which results from interaction between environmental factors and genetic factors. The aim of this study is to investigate the effects of interaction between environmental factors and genetic factors on long-term blood pressure (BP) based on two established cohorts including "the cohort of Hanzhong adolescent hypertension study" and "the cohort of Mei county adult salt-sensitive hypertension study". Firstly, the Hanzhong cohort-based follow-up study is designed to observe the track of BP during the whole life time, and to explore the effects of many risk factors (such as salt-sensitivity, obesity et al) on long-term BP and the occurrence of hypertension, and also to analyze the relationship of different polymorphisms of sodium and potassium metabolism-related gene with BP changes and target organ damages. In addition, by using DNA samples collected from subjects of "Mei county adult salt-sensitive hypertension study"in which all participants had completed a chronic salt loading and potassium intervention trial, we attempt to examine the single nucleotide polymorphisms (SNPs) of sodium and potassium metabolism-related genes, as well as the relationship between these SNPs and BP responses to dietary sodium/potassium intervention, long-term BP change, the risk of hypertension and target organ damages were analyzed. This study would enable us to further explore the etiology of essential hypertension as well as to identify new genetic markers for predicting early hypertension and target organ damage.

DETAILED DESCRIPTION:
This study is a longitudinal cohort follow-up study. The main contents include:(1)Questionnaire design: questionnaire is designed according to the research contents and purposes. The standard questionnaires will be used to collect the general information, dietary habits, lifestyle, medical history and family history etc.(2)Anthropometric measurements: blood pressure, height, body weight,waist and hip, pulse will be acquired by medical practitioners who received professional trainings based on World Health Organization (WHO) standards, and passed relevant examinations.(3) Blood and urine samples collection: morning fasting blood, nocturia, and 24-hour urine specimen will be collected by medical staffs, and blind tubes will be set up according to 5% of the total samples. Blood biochemistries including serum total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides, fasting glucose, creatinine and hsCRP can be measured using automatic biochemical analyzer. The sodium and potassium concentrations in the urine will be measured by flame photometry. The total sodium and potassium excretions in urine in 24h were calculated by multiplying the concentration and 24-h volume of urine. (4) Auxiliary examinations: Auxiliary examinations including carotid intima-media thickness, endothelium-dependent vasodilation (FMD), measurements of brachial-ankle pulse wave velocity (baPWV) and electrocardiographic parameters. The measurement will be done in hospitals by medical practitioners who received professional trainings and passed relevant examinations. (5) Single nucleotide polymorphisms detection: based on our previous studies, sodium and potassium metabolism-related gene polymorphisms will be detected using MassARRAY technology. (6) Data processing and statistics: we should input the data to the database, and utilize softwares such as SPSS, STATA, Haploview and FBAT to analyze. (7) Quality control: ① Questionnaire is strictly designed and amended by epidemiologist and clinical experts. ② A standardized "Investigator Handbook" will be stipulated according to the guidelines. ③ Staff members are required to do a rigorous training and pass the exam. ④ The investigation process will be strictly supervised by the principal investigator. ⑤ Data entry use the parallel double entry method. ⑥ During laboratory testing, blank control and blind detection are applied to ensure the quality. ⑦ Data analysis is performed by 2-3 postgraduates, inconsistent data need to be double checked.

ELIGIBILITY:
Inclusion Criteria:

1. Hanzhong cohort of Adolescent Hypertension Study:

   * adolescents aged 6-15 years old in over 20 schools of three towns (Qili, Laojun and Shayan) in Hanzhong, Shaanxi, China.
2. Mei county cohort of adult salt-sensitive hypertension study:

   * Han individuals in rural northern China
   * adults aged 18-60 years
   * individuals who had a mean systolic BP (SBP) between 130-160 mmHg and/or a diastolic BP (DBP) between 85-100 mmHg and no use of antihypertensive medications were identified as the proband
   * the probands'parents,siblings, spouses, and offspring were recruited for the study.

Exclusion Criteria:

During the follow-up period, the exclusion criteria are as follows:

* Secondary hypertension
* a history of severe cardiovascular disease
* chronic kidney disease or liver disease
* unable to complete the examination
* unable/refuse to sign the informed consent form

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: In March and April, 1987, investigators established the cohort of Hanzhong Adolescent Hypertension Study. A total of 4,623 adolescents aged 6-15 years old in over 20 schools of three towns (Qili, Laojun and Shayan) in Hanzhong, Shaanxi, China were recruited.
  In 2003-2004, investigators established the cohort of Mei county adult salt sensitive hypertension Study. This study was a family-based dietary intervention study conducted in a Han Chinese population from rural areas of northern China. A total of 675 subjects from 126 families were recruited in this cohort.
Sampling Method: Probability Sample
Enrollment: 5298 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
blood pressure value(mmHg) | First day of the three-day follow-up period
  The follow-up study of these two cohorts will last approximately 18 months (Jul 2016 to Dec 2017). During this period, each subject will receive a three-day follow-up examination. Three BP(mmHg) measurements will be obtained using a mercury sphygmomanometer on the first day of the three-day follow-up period.

SECONDARY OUTCOMES:
Left ventricular hypertrophy（g/m^2） | During the three-day follow-up period
  The follow-up study of these two cohorts will last approximately 18 months (Jul 2016 to Dec 2017). During this period, each subject will receive a three-day follow-up examination. Left ventricular mass index (LVMI,g/m^2）will be measured using echocardiography during the three-day follow-up period.
Increased arterial stiffness（mm/s） | During the three-day follow-up period
  The follow-up study of these two cohorts will last approximately 18 months (Jul 2016 to Dec 2017).During this period, each subject will receive a three-day follow-up examination. Brachial-ankle pulse wave velocity（baPWV,mm/s）will be measured with Noninvasive automatic waveform analyzer during the three-day follow-up period.
Carotid artery wall thickening（mm） | During the three-day follow-up period
  The follow-up study of these two cohorts will last approximately 18 months (Jul 2016 to Dec 2017).During this period, each subject will receive a three-day follow-up examination. Carotid Intima media thickness (IMT,mm）will be measured using Color Doppler Ultrasound Diagnostic System during the three-day follow-up period.
Microalbuminuria（mg/24h） | Second day of the three-day follow-up period
  The follow-up study of these two cohorts will last approximately 18 months (Jul 2016 to Dec 2017).During this period, each subject will receive a three-day follow-up examination. On the second day,24-hour urinary will be collected and the concentrations of microalbuminuria in the urine sample will be measured with Hitachi biochemical analyzer.The 24-h microalbuminuria（mg/24h）of each subject is calculated as the concentration of microalbuminuria multiplied by the 24-h urine volume of each individual.

CONTACTS AND LOCATIONS:
Overall Officials: Jianjun Mu, doctor, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
The achievements will be evaluated by papers published in specialized journals with a peer-reviewed system, and the original dates can be disclosed according to requirements.

REFERENCES:
- [Result] Mu J, Zheng S, Lian Q, Liu F, Liu Z. Evolution of blood pressure from adolescents to youth in salt sensitivies: a 18-year follow-up study in Hanzhong children cohort. Nutr J. 2012 Sep 14;11:70. doi: 10.1186/1475-2891-11-70. PMID 22978814
- [Result] Liu F, Zheng S, Mu J, Chu C, Wang L, Wang Y, Xiao H, Wang D, Cao Y, Ren K, Liu E, Yuan Z. Common variation in with no-lysine kinase 1 (WNK1) and blood pressure responses to dietary sodium or potassium interventions- family-based association study. Circ J. 2013;77(1):169-74. doi: 10.1253/circj.cj-12-0900. Epub 2012 Oct 12. PMID 23059770
- [Derived] Wang L, Chang MK, Yue XM, Guo YJ, Yao YN, Liu NR, Yang BB, Niu ZJ, Gao WH, Li H, Wang Y. Associations of Genetic Variations in the NR3C2 With Salt Sensitivity, Longitudinal Blood Pressure Changes, and Incidence of Hypertension in Chinese Adults. J Clin Hypertens (Greenwich). 2025 Sep;27(9):e70137. doi: 10.1111/jch.70137. PMID 40932182
- [Derived] Zhang X, Yao S, Wang Y, Chu C, Du M, Mu J. Associations of microRNA Gene Polymorphisms With Salt Sensitivity, Longitudinal Blood Pressure Changes, and Hypertension Incidence in the Chinese Population. J Clin Hypertens (Greenwich). 2025 Feb;27(2):e70019. doi: 10.1111/jch.70019. PMID 39994918
- [Derived] Liao YY, Wang D, Chu C, Man ZY, Wang Y, Ma Q, Chen C, Sun Y, Mu JJ. Long-term burden and increasing trends of body mass index are linked with adult hypertension through triglyceride-glucose index: A 30-year prospective cohort study. Nutr Metab Cardiovasc Dis. 2024 Sep;34(9):2134-2142. doi: 10.1016/j.numecd.2024.05.014. Epub 2024 May 18. PMID 39003135
- [Derived] Guo T, Zheng S, Chen T, Chu C, Ren J, Sun Y, Wang Y, He M, Yan Y, Jia H, Liao Y, Cao Y, Du M, Wang D, Yuan Z, Wang D, Mu J. The association of long-term trajectories of BMI, its variability, and metabolic syndrome: a 30-year prospective cohort study. EClinicalMedicine. 2024 Feb 12;69:102486. doi: 10.1016/j.eclinm.2024.102486. eCollection 2024 Mar. PMID 38370536
- [Derived] Niu ZJ, Yao S, Zhang X, Mu JJ, Du MF, Zou T, Chu C, Liao YY, Hu GL, Chen C, Wang D, Ma Q, Yan Y, Jia H, Wang KK, Sun Y, Yan RC, Man ZY, Ren DF, Wang L, Gao WH, Li H, Wu YX, Li CH, Gao K, Zhang J, Yang TL, Wang Y. Associations of genetic variations in NEDD4L with salt sensitivity, blood pressure changes and hypertension incidence in Chinese adults. J Clin Hypertens (Greenwich). 2022 Oct;24(10):1381-1389. doi: 10.1111/jch.14566. Epub 2022 Aug 30. PMID 36039789
- [Derived] Yuan Y, Mu JJ, Chu C, Zheng WL, Wang Y, Hu JW, Ma Q, Yan Y, Liao YY, Chen C. Effect of metabolically healthy obesity on the development of arterial stiffness: a prospective cohort study. Nutr Metab (Lond). 2020 Jul 2;17:50. doi: 10.1186/s12986-020-00474-8. eCollection 2020. PMID 32625239
- [Derived] Yuan Y, Chu C, Zheng WL, Ma Q, Hu JW, Wang Y, Yan Y, Liao YY, Mu JJ. Body Mass Index Trajectories in Early Life Is Predictive of Cardiometabolic Risk. J Pediatr. 2020 Apr;219:31-37.e6. doi: 10.1016/j.jpeds.2019.12.060. Epub 2020 Feb 12. PMID 32061408
- [Derived] Yuan Y, Hu JW, Wang Y, Wang KK, Zheng WL, Chu C, Ma Q, Yan Y, Liao YY, Mu JJ. Association between atherogenic index of plasma and subclinical renal damage over a 12-year follow-up: Hanzhong adolescent hypertension study. Eur J Clin Nutr. 2020 Feb;74(2):278-284. doi: 10.1038/s41430-019-0530-x. Epub 2019 Nov 14. PMID 31728032